CLINICAL TRIAL: NCT01904448
Title: An Early Feasibility Study of the Safety and Efficacy of the Nucleus 24 Auditory Brainstem Implant in Children With Cochlear or Cochlear Nerve Disorders Not Resulting From Neurofibromatosis Type II
Brief Title: Auditory Brainstem Implantation in Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-0664
Record Dates: First submitted 2013-07-03; First posted 2013-07-22 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-02

CONDITIONS: Developmental Cochlear Nerve Deficiency; Acquired Cochlear Nerve Deficiency; Cochlear Aplasia; Post-meningitis Cochlear Ossification; Cochlear Malformation
Keywords: pediatric; profound hearing loss; auditory brainstem implant; cochlear implant; developmental or acquired cochlear nerve deficiency (CND); cochlear aplasia (Michel); post-meningitis cochlear ossification; cochlear malformation; CND
MeSH Terms: interventions — Auditory Brain Stem Implantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Auditory Brainstem Implant (Experimental): single-arm study of auditory brainstem implantation in children
  Interventions: Device: Auditory Brainstem Implantation in Children

INTERVENTIONS:
Device: Auditory Brainstem Implantation in Children

SUMMARY:
To purpose of this feasibility study is to demonstrate the safety and efficacy of the Nucleus 24 Multichannel Auditory Brainstem Implant (ABI, Cochlear Corp, Sydney, AUS) in children without the diagnosis of neurofibromatosis type II (NFII) that have either experienced failed cochlear implantation (CI) or have been unable to receive a CI secondary to cochlear or cochlear nerve disorders. These conditions can include: developmental or acquired cochlear nerve deficiency (CND), cochlear aplasia (Michel), post-meningitic cochlear ossification or cochlear malformation.

This study proposes to implant up to 10 young children (<5 yrs. of age) with the Nucleus 24 Multichannel ABI (Sydney, AUS) in an attempt to demonstrate safety of the surgical procedure, tolerance of device stimulation, and the potential for auditory benefit beyond that experienced with their CI. This study will provide the preliminary experience for a larger scale clinical trial.

Aim 1: Demonstrate the safety of ABI surgery in children. Aim 2: Demonstrate the development of sound awareness and improved speech understanding among children implanted with the ABI when compared to their baseline skills. Aim 3: Demonstrate the development of oral language skills following the use of the ABI that were not evident prior to its use.

ELIGIBILITY:
Inclusion Criteria:

* Pre-linguistic hearing loss (birth-5 yrs.; age at ABI 18 months-5yrs) with both:
* MRI +/- CT evidence of one of the following: Cochlear nerve deficiency, Cochlear aplasia or severe hypoplasia, Severe inner ear malformation, Post-meningitis ossification
* When a cochlea is present or patent, lack of significant benefit from CI despite consistent use (>6 mo.)
* Post-linguistic hearing loss (<18 yrs. of age) with both:
* Loss or lack of benefit from appropriate CI without the possibility for revision or contralateral implantation. Examples might include: Post-meningitis ossification, Bilateral temporal bone fractures with cochlear nerve avulsion, Failed revision CI without benefit
* Previously developed open set speech perception and auditory-oral language skills
* No medical contraindications
* Willing to receive the appropriate meningitis vaccinations
* No or limited cognitive/developmental delays which would be expected to interfere with the child's ability to cooperate in testing and/or programming of the device, in developing speech and oral language, or which would make an implant and subsequent emphasis on aural/oral communication not in the child's best interest
* Strong family support including language proficiency of the parent(s) in the child's primary mode of communication as well as written and spoken English.
* Reasonable expectations from parents including a thorough understanding:

  * of potential benefits and limitations of ABI
  * of parental role in rehabilitation
  * that the child may not develop spoken language as a primary communication mode or even sufficient spoken language to make significant academic progress in an aural/oral environment
* Involvement in an educational program that emphasizes development of auditory skills with or without the use of supplementary visual communication.
* Able to comply with study requirements including travel to investigation sites.
* Informed consent for the procedure from the child's parents/legal guardian.

Exclusion Criteria:

* Pre- or post-linguistic child currently making significant progress with CI
* MRI evidence of one of the following:

  * normal cochlea and cochlear nerves or NFII
  * brainstem or cortical anomaly that makes implantation unfeasible
* Clear surgical reason for poor CI performance that can be remediated with revision CI or contralateral surgery rather than ABI.
* Intractable seizures or progressive, deteriorating neurological disorder
* Unable to participate in behavioral testing and mapping with their CI. If this appears to be an age effect, ABI will be delayed until we can be assured that the child will be able to participate, as reliable objective measures of mapping are currently not available for mapping these devices.
* Lack of potential for spoken language development. This will be considered the case when evidence of the following exist:

  * Severe psychomotor retardation, autism, cerebral palsy, or developmental delays beyond speech that would preclude usage of the device and oral educational development. Autism is a special case where there is the potential for delayed presentation. When early signs are considered present, our group routinely requests a comprehensive developmental assessment for further evaluation prior to considering routine evaluation. A specialized group is readily available at our institution for such an evaluation.
* Unable to tolerate general anesthesia (cardiac, pulmonary, bleeding diathesis, etc.).
* Need for brainstem irradiation
* Unrealistic expectations on the part of the subject/family regarding the possible benefits, risks and limitations that are inherent to the procedure and prosthetic device.
* Unwilling to sign the informed consent.
* Unwilling to make necessary follow-up appointments.

Ages: 18 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2012-09; Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig A Buchman, MD, Study Chair — Washington University School of Medicine
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Pediatric Auditory Brainstem Implantation (ABI): Single-arm study of Auditory Brainstem Implantation (ABI) in children
Period: Overall Study
Arm/Group | Pediatric Auditory Brainstem Implantation (ABI)
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Pediatric ABI: Single-arm study of Auditory Brainstem Implantation (ABI) in children
Arm/Group | Pediatric ABI
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 3.4 [2.1 to 5.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of ABI Complications
Description: Complications and related outcomes will be tracked and recorded. These include bleeding, infection, neural injury, cerebrospinal fluid (CSF) leakage, brain bleeding or bruising, stroke, death. Also, complications and sequelae related to the device such as non-auditory stimulation and device failure will be tracked.
Time Frame: Year 3
Measure: Number; unit: Events
Arm/Group | Pediatric ABI
Number analyzed (Participants) | 5
Events | 2

2. Secondary Outcome: The Oral and Written Language Scales (OWLS) Listening Comprehension Score
Description: OWLS-II: Listening Comprehension measures oral language reception, which is the understanding of spoken language. The examiner orally presents increasingly difficult words, phrases, and sentences to the participant and he/she responds by pointing to or stating which of four pictures is correct. The derived mean standard score for this test is 100 with a standard deviation of 15. Higher scores indicate better listening comprehension. Scores of 85 to 115 are within normal limits. Scores that fall 2 standard deviations below the mean are considered to be severely delayed.
Time Frame: Year 3
Measure: Number; unit: units on a scale
Arm/Group | Pediatric ABI
Number analyzed (Participants) | 5
units on a scale
  Subject 1 | 77
  Subject 2 | 46
  Subject 3 | 40
  Subject 4 | 40
  Subject 5 | 62

3. Secondary Outcome: The Oral and Written Language Scales (OWLS) Oral Expression Score
Description: OWLS-II: Oral Expression measures oral language expression, which is the use of spoken language. The examiner presents a verbal prompt along with a picture and the participant must respond orally to the prompt with increasingly difficult language. The derived mean standard score for this test is 100 with a standard deviation of 15. Higher scores indicate better oral expression. Scores of 85 to 115 are within normal limits. Scores that fall 2 standard deviations below the mean are considered to be severely delayed.
Time Frame: Year 3
Measure: Number; unit: units on a scale
Arm/Group | Pediatric ABI
Number analyzed (Participants) | 5
units on a scale
  Subject 1 | 48
  Subject 2 | 50
  Subject 3 | 40
  Subject 4 | 40
  Subject 5 | 58

4. Secondary Outcome: Goldman-Fristoe Test of Articulation Scores (GFTA)
Description: The GFTA-2 is a standardized, norm-based articulation measure that samples spontaneous sound production. Children are asked to respond to picture plates and verbal cues from the examiner with single words that test consonant accuracy in initial, medial, and final positions. This measure has norms based on the performance of normal-hearing children from age 2 years to 21 years.
Time Frame: Year 3
Population: Due to limited progress in spoken language development and test difficulty, this measure was replaced by Identifying Early Phonological Needs in children with hearing loss (IEPN). No data were collected for this measure.
Arm/Group | Pediatric ABI
Number analyzed (Participants) | 0

5. Secondary Outcome: MacArthur-Bates Communicative Development Inventories (CDIs) Score
Description: MacArthur-Bates Communicative Development Inventories (CDIs)
Time Frame: Year 3
Population: Since spoken language skills did not progress as expected, this measure was inappropriate for use in the study and was unobtainable.
Arm/Group | Pediatric ABI
Number analyzed (Participants) | 0

6. Secondary Outcome: Percentage of Correctly Produced Items From the Identifying Early Phonological Needs in Children With Hearing Loss (IEPN) Test-Vocalize on Demand
Description: This is a measure of the child's ability to vocalize on demand elicited by pictures of objects. Scores are derived from the percentage of time the child vocalized for 25 words.
Time Frame: Year 1, Year 2, Year 3
Measure: Number; unit: percentage of correct answers
Arm/Group | Pediatric ABI
Number analyzed (Participants) | 5
percentage of correct answers
  Subject 1 Year 1 | 100
  Subject 1 Year 2 | 100
  Subject 1 Year 3 | 100
  Subject 2 Year 1 | 0
  Subject 2 Year 2 | 100
  Subject 2 Year 3 | 100
  Subject 3 Year 1 | 0
  Subject 3 Year 2 | 0
  Subject 3 Year 3 | 44
  Subject 4 Year 1 | 100
  Subject 4 Year 2 | 100
  Subject 4 Year 3 | 100
  Subject 5 Year 1 | 0
  Subject 5 Year 2 | 0
  Subject 5 Year 3 | 0

7. Secondary Outcome: Percentage of Correctly Produced Items From the Identifying Early Phonological Needs in Children With Hearing Loss (IEPN) Test-Syllables
Description: Measure of percent correct for use of syllables elicited from pictures of single word items. Scores are derived from the percentage of time the child produced the correct number of syllables on 25 items.
Time Frame: Year 1, Year 2, Year 3
Measure: Number; unit: percentage of correct answers
Arm/Group | Pediatric ABI
Number analyzed (Participants) | 5
percentage of correct answers
  Subject 1 Year 1 | 40
  Subject 1 Year 2 | 80
  Subject 1 Year 3 | 92
  Subject 2 Year 1 | 0
  Subject 2 Year 2 | 40
  Subject 2 Year 3 | 80
  Subject 3 Year 1 | 0
  Subject 3 Year 2 | 0
  Subject 3 Year 3 | 40
  Subject 4 Year 1 | 60
  Subject 4 Year 2 | 100
  Subject 4 Year 3 | 60
  Subject 5 Year 1 | 0
  Subject 5 Year 2 | 0
  Subject 5 Year 3 | 0

8. Secondary Outcome: Percentage of Correctly Produced Items From the Identifying Early Phonological Needs in Children With Hearing Loss (IEPN) Test-Initial Consonants
Description: Measure of percent correct on initial consonant production elicited from pictures of single word items. Scores are derived from the percentage of time the child produced an initial consonant on 25 items.
Time Frame: Year 1, Year 2, Year 3
Measure: Number; unit: percentage of correct answers
Arm/Group | Pediatric ABI
Number analyzed (Participants) | 5
percentage of correct answers
  Subject 1 Year 1 | 63
  Subject 1 Year 2 | 95
  Subject 1 Year 3 | 100
  Subject 2 Year 1 | 0
  Subject 2 Year 2 | 66
  Subject 2 Year 3 | 75
  Subject 3 Year 1 | 0
  Subject 3 Year 2 | 0
  Subject 3 Year 3 | 16
  Subject 4 Year 1 | 71
  Subject 4 Year 2 | 38
  Subject 4 Year 3 | 60
  Subject 5 Year 1 | 0
  Subject 5 Year 2 | 0
  Subject 5 Year 3 | 0

9. Secondary Outcome: Percentage of Correctly Produced Items From the Identifying Early Phonological Needs in Children With Hearing Loss (IEPN) Test-Vowels
Description: Measure of percent correct on vowel production elicited from pictures of single word items. Scores are derived from the percentage of time the child produced the correct vowel on 25 items.
Time Frame: Year 1, Year 2, Year 3
Measure: Number; unit: percentage of correct answers
Arm/Group | Pediatric ABI
Number analyzed (Participants) | 5
percentage of correct answers
  Subject 1 Year 1 | 12
  Subject 1 Year 2 | 31
  Subject 1 Year 3 | 53
  Subject 2 Year 1 | 0
  Subject 2 Year 2 | 12
  Subject 2 Year 3 | 26
  Subject 3 Year 1 | 0
  Subject 3 Year 2 | 0
  Subject 3 Year 3 | 20
  Subject 4 Year 1 | 28
  Subject 4 Year 2 | 17
  Subject 4 Year 3 | 45
  Subject 5 Year 1 | 0
  Subject 5 Year 2 | 0
  Subject 5 Year 3 | 0

10. Secondary Outcome: Percentage of Correctly Produced Items From the Identifying Early Phonological Needs in Children With Hearing Loss (IEPN) Test-Manner Cues
Description: Measure of percent correct on consonant manner cues production elicited from pictures of single word items. Scores are derived from the percentage of time the child produced the correct manner of consonant production on 25 items.
Time Frame: Year 1, Year 2, Year 3
Measure: Number; unit: percentage of correct answers
Arm/Group | Pediatric ABI
Number analyzed (Participants) | 5
percentage of correct answers
  Subject 1 Year 1 | 18
  Subject 1 Year 2 | 54
  Subject 1 Year 3 | 56
  Subject 2 Year 1 | 0
  Subject 2 Year 2 | 24
  Subject 2 Year 3 | 24
  Subject 3 Year 1 | 0
  Subject 3 Year 2 | 4
  Subject 3 Year 3 | 4
  Subject 4 Year 1 | 35
  Subject 4 Year 2 | 25
  Subject 4 Year 3 | 37
  Subject 5 Year 1 | 0
  Subject 5 Year 2 | 0
  Subject 5 Year 3 | 0

11. Secondary Outcome: Percentage of Correctly Produced Items From the Identifying Early Phonological Needs in Children With Hearing Loss (IEPN) Test-Final Consonants
Description: Measure of percent correct on final consonant production elicited from pictures of single word items. Scores are derived from the percentage of time the child produced a final consonant on 25 items.
Time Frame: Year 1, Year 2, Year 3
Measure: Number; unit: percentage of correct answers
Arm/Group | Pediatric ABI
Number analyzed (Participants) | 5
percentage of correct answers
  Subject 1 Year 1 | 29
  Subject 1 Year 2 | 64
  Subject 1 Year 3 | 94
  Subject 2 Year 1 | 0
  Subject 2 Year 2 | 0
  Subject 2 Year 3 | 0
  Subject 3 Year 1 | 0
  Subject 3 Year 2 | 0
  Subject 3 Year 3 | 11
  Subject 4 Year 1 | 11
  Subject 4 Year 2 | 41
  Subject 4 Year 3 | 41
  Subject 5 Year 1 | 0
  Subject 5 Year 2 | 0
  Subject 5 Year 3 | 0

12. Secondary Outcome: Percentage of Correctly Produced Items From the Identifying Early Phonological Needs in Children With Hearing Loss (IEPN) Test-Place Cues
Description: Measure of percent correct on consonant place cue production elicited from pictures of single word items. Scores are derived from the percentage of time the child produced the correct place of consonant production on 25 items.
Time Frame: Year 1, Year 2, Year 3
Measure: Number; unit: percentage of correct answers
Arm/Group | Pediatric ABI
Number analyzed (Participants) | 5
percentage of correct answers
  Subject 1 Year 1 | 20
  Subject 1 Year 2 | 58
  Subject 1 Year 3 | 58
  Subject 2 Year 1 | 0
  Subject 2 Year 2 | 27
  Subject 2 Year 3 | 27
  Subject 3 Year 1 | 0
  Subject 3 Year 2 | 0
  Subject 3 Year 3 | 5
  Subject 4 Year 1 | 28
  Subject 4 Year 2 | 21
  Subject 4 Year 3 | 38
  Subject 5 Year 1 | 0
  Subject 5 Year 2 | 0
  Subject 5 Year 3 | 0

13. Secondary Outcome: Percentage of Correctly Produced Items From the Identifying Early Phonological Needs in Children With Hearing Loss (IEPN) Test-Voice Cues
Description: Measure of percent correct on consonant voicing cue production elicited from pictures of single word items. Scores are derived from the percentage of time the child produced the correct voicing of consonant production on 25 items.
Time Frame: Year 1, Year 2, Year 3
Measure: Number; unit: percentage of correct answers
Arm/Group | Pediatric ABI
Number analyzed (Participants) | 5
percentage of correct answers
  Subject 1 Year 1 | 16
  Subject 1 Year 2 | 67
  Subject 1 Year 3 | 90
  Subject 2 Year 1 | 0
  Subject 2 Year 2 | 41
  Subject 2 Year 3 | 25
  Subject 3 Year 1 | 0
  Subject 3 Year 2 | 0
  Subject 3 Year 3 | 3
  Subject 4 Year 1 | 41
  Subject 4 Year 2 | 20
  Subject 4 Year 3 | 51
  Subject 5 Year 1 | 0
  Subject 5 Year 2 | 0
  Subject 5 Year 3 | 0

14. Secondary Outcome: Change in Speech Perception Test Battery Scores-Detection Audiogram
Description: Sound detection for octave frequencies of 250 Hz through 8k Hz were collected and a 4 frequency average was calculated for each annual test interval
Time Frame: Year 1, Year 2, Year 3
Measure: Number; unit: averaged decibel level
Arm/Group | Pediatric ABI
Number analyzed (Participants) | 5
averaged decibel level
  Pure Tone Average (PTA) Subject 1 Year 1 | 30
  PTA Subject 1 Year 2 | 42
  PTA Subject 1 Year 3 | 30
  PTA Subject 2 Year 1 | 120
  PTA Subject 2 Year 2 | 47
  PTA Subject 2 Year 3 | 35
  PTA Subject 3 Year 1 | 33
  PTA Subject 3 Year 2 | 32
  PTA Subject 3 Year 3 | 30
  PTA Subject 4 Year 1 | 32
  PTA Subject 4 Year 2 | 30
  PTA Subject 4 Year 3 | 33
  PTA Subject 5 Year 1 | 35
  PTA Subject 5 Year 2 | 33
  PTA Subject 5 Year 3 | 32

15. Secondary Outcome: Speech Perception Test Battery Scores-IT-MAIS or MAIS
Description: A hierarchy of tests were chosen that capture auditory skills from sound awareness to open set word and sentence understanding. Participants did not advance to the next level of difficulty until demonstrating a minimum performance on the previous measure.
  The Infant-Toddler Meaningful Auditory Integration Scale (IT-MAIS) is a parent questionnaire consisting of ten questions regarding a young infant or toddler's auditory behavior, e.g., "Does the child spontaneously respond to his/her name in quiet with auditory cues?" Each question is scored on a five point scale: 0 = never, 1 = rarely, 2 = occasionally, 3 = frequently, and 4 = always. The aim of this tool is to assess the benefit of the child's personal amplification device(s) and is used to assess hearing aid benefit. Higher scores reflect more consistent auditory response. Scores reported are the percentage of correctly answered questions of the total asked.
Time Frame: Pre-ABI, Year 1, Year 2, Year 3
Measure: Number; unit: percent correct
Arm/Group | Pediatric ABI
Number analyzed (Participants) | 5
percent correct
  Subject 1 Pre-ABI | 3
  Subject 1 Year 1 | 43
  Subject 1 Year 2 | 32
  Subject 1 Year 3 | 42
  Subject 2 Pre-ABI | 0
  Subject 2 Year 1 | 28
  Subject 2 Year 2 | 12
  Subject 2 Year 3 | 72
  Subject 3 Pre-ABI | 0
  Subject 3 Year 1 | 52
  Subject 3 Year 2 | 70
  Subject 3 Year 3 | 33
  Subject 4 Pre-ABI | 75
  Subject 4 Year 1 | 50
  Subject 4 Year 2 | 55
  Subject 4 Year 3 | 52
  Subject 5 Pre-ABI | 0
  Subject 5 Year 1 | 2
  Subject 5 Year 2 | 5
  Subject 5 Year 3 | 0

16. Secondary Outcome: Change in Speech Perception Test Battery Scores-Ling Sound Test
Description: A hierarchy of tests were chosen that capture auditory skills from sound awareness to open set word and sentence understanding. Participants did not advance to the next level of difficulty until they demonstrated a minimum performance on the previous measure.
  The Ling- 6 sounds test is a speech sound detection measurement of detection thresholds performed by an audiologist. Six sound files of "ah", "ee", "oo", "sh", "s", and "m" are presented one at a time in varying order for measurement of hearing threshold groups, per sound. The selected sounds tested validate hearing device fitting across the frequency range important for understanding speech. If the child can detect the stimuli a point is given and if they can not detect, no point is given. A total of 3 trials per sound were presented for a total of 18 presentations. The score reflects a percent of the total sounds that were detected.
Time Frame: Year 1, Year 2, Year 3
Population: Single-arm study of Auditory Brainstem Implantation (ABI) in children
Measure: Number; unit: percent correct
Arm/Group | Pediatric ABI
Number analyzed (Participants) | 5
percent correct
  Ling 6 Subject 1 Year 1 | 100
  Ling 6 Subject 1 Year 2 | 100
  Ling 6 Subject 1 Year 3 | 100
  Ling 6 Subject 2 Year 1 | 0
  Ling 6 Subject 2 Year 2 | 100
  Ling 6 Subject 2 Year 3 | 100
  Ling 6 Subject 3 Year 1 | 100
  Ling 6 Subject 3 Year 2 | 100
  Ling 6 Subject 3 Year 3 | 100
  Ling 6 Subject 4 Year 1 | 100
  Ling 6 Subject 4 Year 2 | 100
  Ling 6 Subject 4 Year 3 | 100
  Ling 6 Subject 5 Year 1 | 100
  Ling 6 Subject 5 Year 2 | 100
  Ling 6 Subject 5 Year 3 | 100

17. Secondary Outcome: Change in Speech Perception Test Battery Scores-ESP Low Verbal
Description: A hierarchy of tests were chosen that capture auditory skills from sound awareness to open set word and sentence understanding. Participants did not advance to the next level of difficulty until they demonstrated a minimum performance on the previous measure.
  The Early Speech Perception (ESP) low verbal version estimates speech perception abilities in very young children who have limited verbal abilities. Stimuli consist of words varying in pattern as well as spondees and monosyllabic words presented in sets of four. The format is four item closed-set. Test materials consist of objects (toys) instead of pictures. It is scored by the percent of correctly identified items from the set of 4; 3 repetitions of each item are given for a total of 12 trials.
Time Frame: Year 1, Year 2, Year 3
Population: Missing values indicate test was not administered at that interval and ESP-Standard was administered.
Measure: Number; unit: percentage of correct answers
Arm/Group | Pediatric ABI
Number analyzed (Participants) | 4
percentage of correct answers
  Pattern Subject 1 Year 1 | 25
  Monosyllable Subject 1 Year 1 | 58
  Spondee Subject 1 Year 1 | 25
  Pattern Subject 1 Year 2 | 100
  Monosyllable Subject 1 Year 2 | 75
  Spondee Subject 1 Year 2 | 67
  Pattern Subject 2 Year 1 | 25
  Monosyllable Subject 2 Year 1 | 25
  Spondee Subject 2 Year 1 | 25
  Pattern Subject 2 Year 2 | 25
  Monosyllable Subject 2 Year 2 | 25
  Spondee Subject 2 Year 2 | 25
  Pattern Subject 2 Year 3 | 25
  Monosyllable Subject 2 Year 3 | 25
  Spondee Subject 2 Year 3 | 25
  Pattern Subject 3 Year 1 | 25
  Monosyllable Subject 3 Year 1 | 25
  Spondee Subject 3 Year 1 | 25
  Pattern Subject 3 Year 2 | 83
  Monosyllable Subject 3 Year 2 | 25
  Spondee Subject 3 Year 2 | 25
  Pattern Subject 5 Year 1 | 25
  Monosyllable Subject 5 Year 1 | 25
  Spondee Subject 5 Year 1 | 25
  Pattern Subject 5 Year 2 | 25
  Monosyllable Subject 5 Year 2 | 25
  Spondee Subject 5 Year 2 | 25
  Pattern Subject 5 Year 3 | 25
  Monosyllable Subject 5 Year 3 | 25
  Spondee Subject 5 Year 3 | 25

18. Secondary Outcome: Change in Speech Perception Test Battery Scores-ESP Standard
Description: A hierarchy of tests were chosen that capture auditory skills from sound awareness to open set word and sentence understanding. Participants did not advance to the next level of difficulty until they demonstrated a minimum performance on the previous measure. This may have been due to child's age or inability to complete task. The Early Speech Perception (ESP) Standard measures the progression of speech discrimination skills in children (age 5+) with profound hearing loss as they develop. The stimuli consist of 3 subtests [1) patterns and words, 2) monosyllable, 3) spondees] of 12 pictured words each presented in an auditory-only condition. The format is a closed-set. Two repetitions of each item are given for a total of 24 items for each subtest. Each subtest is scored by the percent of correctly identified items from the set of pictured words.
Time Frame: Year 1, Year 2, Year 3
Population: Missing values indicate test was not administered at that interval and ESP-LV (Low Verbal) was administered.
Measure: Number; unit: percentage of correct answers
Arm/Group | Pediatric ABI
Number analyzed (Participants) | 3
percentage of correct answers
  Pattern Subject 1 Year 3 | 70
  Word Subject 1 Year 3 | 62
  Monosyllable Subject 1 Year 3 | 50
  Spondee Subject 1 Year 3 | 41
  Pattern Subject 3 Year 2 | 66
  Word Subject 3 Year 2 | 41
  Monosyllable Subject 3 Year 2 | 25
  Spondee Subject 3 Year 2 | 25
  Pattern Subject 3 Year 3 | 46
  Word Subject 3 Year 3 | 29
  Monosyllable Subject 3 Year 3 | 25
  Spondee Subject 3 Year 3 | 25
  Pattern Subject 4 Year 1 | 50
  Word Subject 4 Year 1 | 45
  Monosyllable Subject 4 Year 1 | 25
  Spondee Subject 4 Year 1 | 25
  Pattern Subject 4 Year 2 | 45
  Word Subject 4 Year 2 | 41
  Monosyllable Subject 4 Year 2 | 16
  Spondee Subject 4 Year 2 | 25
  Pattern Subject 4 Year 3 | 53
  Word Subject 4 Year 3 | 42
  Monosyllable Subject 4 Year 3 | 8
  Spondee Subject 4 Year 3 | 42

19. Secondary Outcome: Pre-School Language Scale (PLS-5) Scores
Description: The PLS-5 is a standardized language test designed for infants and young children. The Auditory Comprehension subscale targets skills known to precede language development, including: attention to speakers, appropriate object play, basic vocabulary, concepts, grammatical markers, and complex sentences. The Expressive Communication subscale assesses vocal development, social communication, naming of common objects, phonological awareness, sequencing skills, as well as use of concepts, prepositions, grammatical markers, and varying sentence structures.
Time Frame: Year 1, Year 2, Year 3
Population: as for outcome 5
Arm/Group | Pediatric ABI
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the three year study course following enrollment for each participant.
Arm/Group | Pediatric ABI
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pediatric ABI (N=5)
Cerebral Spinal Fluid (CSF) Leak (Surgical and medical procedures) | 1 (1) — CSF wound leakage requiring second surgery to reinforce close and placement of lumbar drain.
Aseptic Meningitis (Surgical and medical procedures) | 1 (1) — Presumptive diagnosis of bacterial meningitis although negative gram stain and cultures throughout. Treated with six weeks of IV antibiotics with resolution.

LIMITATIONS AND CAVEATS:
This study included only 5 participants and statistically reliable results were not possible. There was a floor effect for measures chosen to demonstrate device efficacy; they were found to be unspecific and insensitive to change observed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-06-30): https://cdn.clinicaltrials.gov/large-docs/48/NCT01904448/Prot_SAP_000.pdf